CLINICAL TRIAL: NCT01708473
Title: Feasibility Study: Comparison Of Advil® Vs. Lortab® For Reducing Discomfort Associated With Ultherapy™ Treatment
Brief Title: Feasibility Study: Compare the Effectiveness Between Two Pain Medications When Used Prior to Ultherapy™ Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ULT-123
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-06

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa | interventions — Ibuprofen; oxycodone-acetaminophen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Advil with Ultherapy (Active Comparator): Subjects randomized to this study arm will receive Advil prior to an Ulthera System Treatment.
  Interventions: Drug: Advil; Device: Ulthera System Treatment
- Lortab with Ultherapy (Active Comparator): Subjects randomized to this study arm will receive Lortab prior to an Ulthera System Treatment.
  Interventions: Drug: Lortab; Device: Ulthera System Treatment

INTERVENTIONS:
Drug: Advil — One (1) tablet 800 mg Advil one hour prior to treatment.
  Arms: Advil with Ultherapy
Drug: Lortab — One (1) tablet 10/500 mg of Lortab one hour prior to treatment.
  Arms: Lortab with Ultherapy
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening

SUMMARY:
This study will compare the effectiveness of two pain medications for reducing discomfort during an Ultherapy treatment.

DETAILED DESCRIPTION:
This trial is a prospective, single-site, double-blinded, randomized trial. All study subjects will receive a full face and neck Ultherapy treatment. Subjects will be randomized to receive one of two pain medications prior to treatment. Each subject will be asked to rate the level of discomfort during the Ultherapy treatment. All study subjects will be followed for 90 days following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 30 to 65 years
* Subject in good health
* Skin laxity on the upper and lower face and neck
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the followup period

Exclusion Criteria:

* Known sensitivity to ibuprofen, acetaminophen, or opiates
* Presence of an active systemic or local skin disease that may affect wound healing
* Severe solar elastosis
* Excessive subcutaneous fat in the face and neck
* Excessive skin laxity on the face and neck
* Significant scarring in areas to be treated
* Significant open facial wounds or lesions
* Severe or cystic acne on the face
* Presence of a metal stent or implant in the facial area to be treated

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Treatment discomfort | During treatment
  The validated NRS scale will be used to measure average pain scores reported by subject during treatment.

SECONDARY OUTCOMES:
Improvement in skin laxity | 90 days following treatment
  Improvement in overall lifting and tightening of skin as determined by a masked, qualitative assessment of photographs.

CONTACTS AND LOCATIONS:
Overall Officials: Hema Sundaram, MD, Principal Investigator — Dermatology, Cosmetic & Laser Surgery
Locations (1):
- Dermatology, Cosmetic & Laser Surgery, Rockville, Maryland, United States